CLINICAL TRIAL: NCT05184881
Title: Comparison Between Retrolaminar and Medial Branch Block in Cervical Facet Joint Arthropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, assist. prof. of anesthesia and pain management, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.21.11.1534
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Joint Pain
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group medial branch block (Active Comparator): cervical medial branch block will done at the affected dermatomal level using 1 mL of a mixture of 0.5 mL 1% lidocaine and 0.5 mL dexamethasome (8mg/2ml).
  Interventions: Other: Medial Branch Block
- Group retrolaminar block (Active Comparator): cervical retrolaminar block was done using 5 mL of a mixture of 3 mL 1% lidocaine and 2 mL dexamethasome (8mg/2ml) for each affected dermatomal level.
  Interventions: Other: Retrolaminar block

INTERVENTIONS:
Other: Retrolaminar block — 2- Cervical retrolaminar block: will be performed on prone-positioned patients. Under fluoroscopic visualization, after identification of the lamina at the desired level, a 25-gauge, 3.5-inch spinal needle was introduced and when the needle tip will be confirmed at the posterior aspect of the cervical lamina corresponding to cervical facet arthropathy level. 5 mL of a mixture of 3 mL 1% lidocaine and 2 mL dexamethasome (8mg/2ml) will be injected.
  Arms: Group retrolaminar block
Other: Medial Branch Block — 1- Cervical medial branch block: will be performed on prone-positioned patients using a posterior approach. Under fluoroscopic visualization, after identification of the waists of the articular pillars at the desired levels, each medial branch block was administered with a 25-gauge, 3.5-inch spinal needle. When the place of the needle tip will be confirmed at the mid-point of the waists of articular pillars, 1 ml of the mixture of 0.5 mL 1% lidocaine and 0.5 mL dexamethasome (8mg/2ml) will be injected at each level.
  Arms: Group medial branch block

SUMMARY:
Cervical facet joints have been implicated as a source of chronic pain in 54-67 % patients with chronic posterior neck pain.1 Intraarticular injections, medial branch nerve blocks and neurolysis of medial branch nerves have been described in managing chronic neck pain of facet joint origin.2 The evidence for long-term therapeutic benefits of intraarticular injections of facet joints is limited. Medial branch nerve blocks show moderate evidence of long-term benefit with evidence of side effects.3 Paraneuraxial nerve blocks have become very popular clinically, due to their clinical and anatomical characteristics. These techniques are comparable to neuraxial nerve blocks in terms of success rate and analgesic efficacy and may confer many of advantages over neuraxial nerve blocks.4 Retrolaminar blocks are among this family that are near but not within the neuraxis like spinals or epidurals.5 Most reports and studies of retrolaminar blocks have been in the context of anesthesia for truncal surgery and truncal pain syndromes (thoracic and abdominal).6 Postoperative and pain treatment cervical retrolaminar blocks studies are currently sparse.7 The major advantage of this technique is minimizing or even eliminating the risk of pneumothorax. Additionally, the risks of nerve root damage and inadvertent injection into a dural sleeve, an intervertebral foramen, or the epidural or intrathecal spaces should also be decreased.8

DETAILED DESCRIPTION:
This prospective randomized open comparative study will be conducted in pain clinic, Mansoura University Hospitals. The study will be approved by the Ethics Research Committee of the Faculty of Medicine, Mansoura University and will be carried out in compliance with the Helsinki Declaration. Informed written consent will be signed from every patient participating in this study after full description of all details of every aspect in this study.

The study participants were randomly grouped on a scale of 1:1, using a computer-generated list of random numbers. The distribution results were sealed in an opaque envelope and kept by the study administrator. On the day of block, the study manager handed the envelope to the anesthesiologist who will perform the block.

Grouping:

* Group M: cervical medial branch block will done at the affected dermatomal level using 1 mL of a mixture of 0.5 mL 1% lidocaine and 0.5 mL dexamethasome (8mg/2ml).
* Group R: cervical retrolaminar block was done using 5 mL of a mixture of 3 mL 1% lidocaine and 2 mL dexamethasome (8mg/2ml) for each affected dermatomal level.

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years old of both genders with cervical facet joint arthropathy confirmed by magnetic resonance imaging (MRI) and neck manual examination and not responding to conservative treatments
* numeric rating scale (NRS) ≥ 4 that ranged from 0 (no pain) to 10 (extreme pain).,
* American society of Anesthesiology Physical Status class I and II,
* Body mass index ˂ 30

Exclusion Criteria:

* The exclusion criteria are patient refusal
* local or systemic sepsis, coagulopathy,
* unstable cardiovascular and respiratory diseases,
* previous neurological deficits,
* history of psychiatric disorders,
* history of drug abuse,
* distorted local anatomy,
* those who were allergic to the used medications .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Numerical rating score | before injection
  from zero to 10 (where 0 no pain, 10 the worst pain)
Numerical rating score | after 2 weeks from injection
  from zero to 10 (where 0 no pain, 10 the worst pain)
Numerical rating score | after 2 month from block
  from zero to 10 (where 0 no pain, 10 the worst pain)
Numerical rating score | after 3 month from block
  from zero to 10 (where 0 no pain, 10 the worst pain)

SECONDARY OUTCOMES:
Neck disability index | before injection
  Each of the 10 items scores from 0 to 5. The maximum score is 50. 0 to 4 = no disability, 5 to 14 = mild, 15 to 24 = moderate, 25 to 34 = severe and above 34 = complete.
Neck disability index | after 2 weeks from injection
  Each of the 10 items scores from 0 to 5. The maximum score is 50. 0 to 4 = no disability, 5 to 14 = mild, 15 to 24 = moderate, 25 to 34 = severe and above 34 = complete.

CONTACTS AND LOCATIONS:
Locations (1):
- Yahya Wahba, Al Mansurah, Egypt